CLINICAL TRIAL: NCT02163850
Title: SALUS Trial TranScatheter Aortic Valve RepLacement System Pivotal Trial The Safety and Effectiveness of the Direct Flow Medical Tanscatheter Aortic Valve System
Brief Title: Transcatheter Aortic Valve Replacement System Pivotal Trial
Acronym: SALUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direct Flow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP 011, G120160
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct Flow Medical (Experimental): Direct Flow Medical Transcatheter Aortic Valve Replacement System (TAVR)
  Interventions: Device: Direct Flow Medical
- Commercially Available (Active Comparator): Medtronic CoreValve Transcatheter Aortic Valve Replacement System (TAVR) or Edwards SAPIEN Transcatheter Aortic Valve Replacement System (TAVR)
  Interventions: Device: Commercially Available

INTERVENTIONS:
Device: Direct Flow Medical — Direct Flow Medical Transcatheter Aortic Valve Replacement System (TAVR)
  Other Names: TAVR
  Arms: Direct Flow Medical
Device: Commercially Available — Medtronic CoreValve Transcatheter Aortic Valve Replacement System (TAVR) or Edwards SAPIEN Transcatheter Aortic Valve Replacement System (TAVR)
  Other Names: TAVR
  Arms: Commercially Available

SUMMARY:
Prospective, randomized, unblinded, multi-center investigational study with enrollment at up to 45 investigational sites. The study is designed to compare the study device (Direct Flow Medical Transcatheter Aortic Valve System) composite event rate to a blended commercial comparator (using approved Medtronic self-expanding bioprosthesis or Edwards balloon-expandable bioprosthesis) in high and extreme risk Subjects with severe symptomatic aortic stenosis. Subjects will be followed through the index procedure, hospital discharge, and at 30 days, 6 months and 1 year for the primary endpoint analysis. Thereafter, annual follow-up at 2 through 5 years will be conducted and analyzed separately.

DETAILED DESCRIPTION:
Prospective, randomized, unblinded, multi-center investigational study with enrollment at up to 45 investigational sites. The study is designed to compare the study device (Direct Flow Medical Transcatheter Aortic Valve System) composite event rate to a blended commercial comparator (using approved Medtronic self-expanding bioprosthesis or Edwards balloon-expandable bioprosthesis) in high and extreme risk Subjects with severe symptomatic aortic stenosis. Subjects will be followed through the index procedure, hospital discharge, and at 30 days, 6 months and 1 year for the primary endpoint analysis. Thereafter, annual follow-up at 2 through 5 years will be conducted and analyzed separately.

The primary study endpoint is a composite of all-cause mortality, disabling stroke, or moderate or greater residual aortic regurgitation (based on core lab assessment) at 1 year. All primary endpoint events will be evaluated by a CEC using the definitions located in this protocol.

A sample size of 648 subjects (432 subjects in Direct Flow Medical Transcatheter Aortic Valve System cohort + 216 subjects in blended control cohort) will provide at least 85% power to test that the study device is non-inferior to the comparator with non-inferiority margin of 10%.

Subjects must meet the fundamental enrollment criteria of severe symptomatic, calcific aortic stenosis with quantifiable and documented source records.

ELIGIBILITY:
Inclusion criteria:

1. The subject has severe senile degenerative aortic valve stenosis determined by echocardiogram and Doppler, or simultaneous pressure recordings at cardiac catheterization defined as: mean aortic gradient ≥40 mmHg, or an aortic valve area ≤1.0 cm2 or aortic valve area index ≤0.6 cm2/m2.
2. The subject has moderate to severe symptoms from aortic valve stenosis (NYHA Functional Class ≥II).
3. Subject has a documented aortic annulus size of ≥22 mm and <29 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Patient Review Committee [PRC]) and is deemed treatable with an available size of both test and control device.
4. There is agreement by the heart team (which must include a site cardiac interventionalist and two cardiac surgeons which can be either two cardiac surgeon staff members at the hospital where the procedure is to be performed or one surgeon from the hospital where the procedure is to be performed and a surgeon from the referring institution or practice) that subject is at high operative risk or greater of serious morbidity or mortality with surgical valve replacement (see note below for definitions of extreme and high risk, the required level of surgical assessment, and PRC confirmation) and that TAVR is appropriate. Subjects will be designated either extreme risk (defined as a mortality or irreversible morbidity 50% or great at 30 days) or high risk (i.e., Society of Thoracic Surgeons operative risk score >8% or at a > 15% risk of surgical mortality at 30 days but not extreme risk). This conclusion shall be based on consensus of one cardiac interventionalist and two cardiac surgeons that have reviewed the case after careful consideration of the Subject's STS risk score and co-morbidities.
5. Subject understands the study requirements and the treatment procedures, and provides written informed consent.
6. Subject agrees and is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion criteria:

1. Left ventricular ejection fraction (LVEF) <20% determined by resting echocardiogram.
2. Subjects with an acute STEMI within 30 days preceding the index procedure.
3. Chronic kidney disease with creatinine clearance < 20 ml/min.
4. Subjects with a platelet count of <50,000 cells/mm³ or a WBC < 1000 cells/mm³ within 7 days prior to index procedure.
5. Subject has a known contraindication or hypersensitivity to all antithrombin regimens (aspirin, all P2Y12 inhibitors) that cannot be adequately pretreated, or inability to be anti-coagulated for the study procedure. Note: Subjects who require chronic anticoagulation must be able to be treated additionally with either aspirin or clopidogrel.
6. Any subject with a balloon valvuloplasty (BAV) within 72 hours prior to the index procedure.
7. Subjects who are on a waiting list for any organ transplant.
8. Subjects with known other medical illness associated with a life expectancy of less than one year, or expectation that subject will not improve despite treatment of aortic stenosis.
9. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to nickel, tantalum, titanium, or polyurethanes.
10. Subjects with a history of a stroke or transient ischemic attack (TIA) within previous 60 days of index procedure.
11. Subjects with an active gastrointestinal (GI) bleed or bleeding precluding dual antiplatelet therapy.
12. Subjects presenting with hemodynamic instability or cardiogenic shock requiring inotropic support or mechanical support devices.
13. Subjects who have a planned treatment with any other investigational device or procedure through 1 year follow-up, or who are currently participating in an investigational drug or another device trial.
14. Any planned surgical, percutaneous coronary or peripheral procedure to be performed within the 30 day follow-up from the TAVR procedure.
15. Untreated clinically significant coronary artery disease requiring revascularization.
16. Newly identified left atrial thrombus that has not been treated.
17. Active endocarditis or sepsis within 6 months prior to the study procedure.
18. Any condition resulting in inability to provide informed consent for the trial or difficulty in assessment of neurologic status.
19. Congenital bicuspid or unicuspid valve.
20. Prior aortic valve surgery or pre-existing prosthetic heart valve in any position (mitral and tricuspid rings are permissible).
21. A native valve annulus diameter <22mm or >29mm determined by the screening CT scan.
22. Echocardiographic evidence of new intra-cardiac mass, untreated thrombus, or vegetation that requires treatment.
23. >3+: aortic regurgitation, mitral regurgitation or tricuspid regurgitation.
24. Severe mitral or tricuspid stenosis.
25. Thoracic aortic aneurysm (TAA) >5.50 cm.
26. Inability to transfuse blood.
27. Subject has femoral arterial access that is not acceptable for the study as defined in the device Instructions for Use.
28. Coronary anatomy that precludes the perfusion of native coronary arteries post-implant.
29. Prohibitive left ventricular outflow tract (LVOT) calcification that would prevent proper deployment of a transcatheter valve.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 878 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Death (all cause) and disabling stroke. | 12 Months
  The primary study endpoint is a composite of all-cause mortality, disabling stroke, or moderate or greater residual aortic regurgitation (based on core lab assessment) at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lim, M.D., Principal Investigator — Associate Professor of Pediatrics and Medicine and Director of Advanced Cardiac Valve Center at University of Virginia; Isacc George, Principal Investigator — Columbia University, Assitant Professor of Surgery Division of Cadiothoracic Surgery
Locations (3):
- United States (3):
  - NewYork-Presbyterian / Columbia Univ., New York, New York
  - Ohio Health Riverside Methodist, Columbus, Ohio
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided